CLINICAL TRIAL: NCT06904235
Title: A Multicentre, Multinational, Pharmacokinetic, Safety, and Efficacy Study With IV NEPA (Fosnetupitant/Palonosetron) for the Prevention of Chemotherapy-induced Nausea and Vomiting in Paediatric Cancer Patients Undergoing Highly Emetogenic Chemotherapy (HEC). A 2-part Study With Phase 2, Open-label, Randomised, Single-dose IV NEPA vs Fosaprepitant/Ondansetron in Single-day HEC and Repeated-dose IV NEPA in Multi-day HEC (Part I, Single Cycle) and With Phase 3, Double-blind, Randomised, Repeated-dose IV NEPA vs Fosaprepitant/Ondansetron in Multi-day HEC (Part II, Repeated Cycles)
Brief Title: Study With IV NEPA (Fosnetupitant/Palonosetron) for the Prevention of Chemotherapy-induced Nausea and Vomiting in Paediatric Cancer Patients Undergoing Highly Emetogenic Chemotherapy (HEC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NEPA-22-01; 2024-514321-39 (EudraCT Number)
Record Dates: First submitted 2024-12-16; First posted 2025-04-01 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Nausea and Vomiting Chemotherapy-Induced; Nausea Post Chemotherapy
Keywords: Prevention of chemotherapy-induced nausea and vomiting; highly emetogenic chemotherapy; HEC; IV NEPA; CINV
MeSH Terms: conditions — Nausea; Vomiting | interventions — Palonosetron

STUDY DESIGN:
Intervention Model Description: * Cohort 1: Single-day HEC and single-dose administration of Test Treatment (IV NEPA) or administration of Reference Treatment (IV fosaprepitant + IV ondansetron) on Day 1. Due to fosaprepitant and ondansetron not being indicated in patients younger than 6 months of age and due to fosaprepitant not being indicated in patients with body weight <6 kg, in Cohort 1, patients aged <6 months will exclusively receive the Test Treatment. Patients aged ≥6 months and weighing at least 6 kg will be randomly allocated to either Test Treatment or Reference Treatment.
  * Cohort 2: Multi-day HEC and repeated-dose administration of Test Treatment (IV NEPA), with the first administration on Day 1. All patients will receive the Test Treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV NEPA (Experimental): The Test Treatment (IV NEPA) is planned to be administered in Cohort 1 and Cohort 2.
  IV NEPA Dosing Schedule
  * Cohort 1 (single-day HEC): Single 30-min infusion on Day 1, before start of chemotherapy.
  * Cohort 2 (multi-day HEC): Single 30-min infusion on Days 1, 3, and 5 (administration on Day 5 depending on the patient's multi day HEC scheme), before start of chemotherapy or in the morning if no chemotherapy is administered on the same day.
  Interventions: Drug: IV NEPA (fosnetupitant/palonosetron)
- Reference Treatment (Active Comparator): The Reference Treatment is planned to be administered in Cohort 1 only. The Reference Treatment includes fosaprepitant powder for solution for IV infusion and ondansetron liquid solution for IV infusion.
  Interventions: Drug: Reference Treatment: IV ondansetron infusion; Drug: Reference Treatment: IV fosaprepitant infusion

INTERVENTIONS:
Drug: IV NEPA (fosnetupitant/palonosetron) — In NEPA-22-01, different body weight-based dosages of IV NEPA will be applied to patients below and over 3 months of age:
  Formulation A (for patients ≥3 months of age; 235 mg fosnetupitant/1.5 mg palonosetron per vial) or Formulation B (for patients <3 months of age; 235 mg fosnetupitant/2.5 mg palonosetron per vial).
  Arms: IV NEPA
Drug: Reference Treatment: IV ondansetron infusion — IV Ondansetron Dosing Regimen
  * Day 1 (before start of chemotherapy): One 30-min infusion of 0.15 mg/kg (ondansetron maximum dose: 8 mg per administration)
  * Day 1 at 4 h and 8 h after the end of first administration: Two 30-min infusions of 0.15 mg/kg (ondansetron maximum dose: 8 mg per administration)
  Arms: Reference Treatment
Drug: Reference Treatment: IV fosaprepitant infusion — Fosaprepitant IV Dosing Regimen
  * Patients aged 12 years to <18 years: a single dose of IV fosaprepitant 150 mg
  * Patients aged 2 years to <12 years: a single dose of IV fosaprepitant 4 mg/kg (maximum dose: 150 mg)
  * Patients aged 6 months to <2 years: a single dose of IV fosaprepitant 5 mg/kg (maximum dose: 150 mg)
  Arms: Reference Treatment

SUMMARY:
Chemotherapy often causes nausea and vomiting (CINV), and this is a major problem for the children being treated for cancer. To prevent this, a combination of two substances in fixed proportion (IV NEPA) was developed. The two substances are: palonosetron, an antagonist of 5 HT3 receptors, and fosnetupitant, an antagonist of NK1 receptors that transforms into netupitant in the body. The medication is administered through intravenous injection (IV- drip).

This study is built from 2 parts:

Part 1: phase 2, open label Part 2: phase 3 double blind

The detailed description, study design, study milestones and eligibility criteria will reflect the Part 1 requirements

DETAILED DESCRIPTION:
Part I of the study is a Phase 2, open-label, randomised (for Cohort 1 only), single chemotherapy cycle study which will compare single-dose of IV NEPA to another treatment (fosaprepitant/ondansetron) considered as a standard of care, in patients receiving single-day chemotherapy that has a high possibility to generate a vomiting episode (HEC) (Cohort 1) and assess repeated dose of IV NEPA in patients receiving multi day HEC chemotherapy (Cohort 2).

Because this will be the first study testing the IV NEPA in children, Part I will enroll patients from older to younger age groups with safety checks before moving to the next group.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria must be checked prior to study inclusion:

1. Signed written Informed Consent Form (ICF) by parent(s)/legal guardian of the paediatric patient in compliance with the local laws and regulations. In addition, the signed children's Assent Form according to local requirements.
2. Male or female in- or out-patient from 0 months (newborns) to <18 years on the date of enrolment (Day 1).
3. Cohort 1: Patient < 6 months weighing at least 4 kg or patient ≥ 6 months weighing at least 6 kg.

   Cohort 2: Patient weighing at least 4 kg.
4. Patient with a predicted life expectancy ≥3 months according to Investigator's opinion.
5. Patient naïve or non-naïve to chemotherapy, with histologically and/or cytologically (or imaging in the case of brain tumours and nephroblastomas) confirmed malignant disease.
6. Cohort 1: Patient scheduled and eligible to receive at least 1 cycle of single-day HEC.

   Cohort 2: Patient scheduled and eligible to receive at least 1 cycle of multi-day HEC.

   (For the level of emetogenicity of the chemotherapeutic agents, refer to the POGO January 2021 guideline).
7. For patients aged ≥10 years: Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤2.
8. For patient with known hepatic impairment: the patient may be enrolled provided the serum ALT and AST are ≤2.5 ULN, the total bilirubin is ≤1.5 ULN, and in the Investigator's opinion the impairment is not expected to jeopardize the patient's safety during the study.
9. For patient with known renal impairment: the patient may be enrolled provided the estimated glomerular filtration rate (eGFR) is ≥70 mL/min/1.73m2 (≥50 mL/min/1.73m2 for children <3 months old) (the eGFR should be calculated using the modified Schwartz equation) and in the Investigator's opinion the impairment is not expected to jeopardize the patient's safety during the study.
10. For patient with known history or predisposition to cardiac abnormalities: as per the Investigator's opinion, the history/predisposition should not jeopardize patient's safety during the study.
11. Patient with non-clinically significant abnormal laboratory values or with clinically relevant abnormal laboratory values may be enrolled if in the Investigator's opinion the patient's safety is not expected to be jeopardized.
12. Female patient shall: a) not have attained menarche yet or b) have attained menarche and have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at Day 1.
13. Male or female fertile patient using reliable contraceptive measures. Such measures, for patient and sexual partner, include: implants, injectables, combined oral contraceptives, intrauterine devices, vasectomized/sterilized partner, use of a double barrier method, or sexual abstinence. The patient and his/her parent(s)/legal guardian must be counselled on the importance of avoiding pregnancy before and during the study.

Exclusion Criteria:

1. The patient and/or parent(s)/legal guardian are expected by the Investigator to be non compliant with the study procedures.
2. Patient has received or is scheduled to receive total body irradiation; total nodal irradiation; upper abdomen radiotherapy; half or upper body irradiation; or radiotherapy of the cranium, craniospinal regions, head and neck, lower thorax region, or the pelvis within 1 week prior to study entry (Day 1) or within 120 h after start of chemotherapy on Day 1 (Cohort 1 patients) or within 168 h (for Cohort 2 patients receiving the last IV NEPA on Day 3) or 216 h (for Cohort 2 patients receiving the last IV NEPA on Day 5) from start of chemotherapy on Day 1.
3. Known history of allergy to any component of the study treatments or other contraindications to any NK1-RAs or 5-HT3-RAs.
4. Active infection.
5. Any illness or condition that, in the opinion of the Investigator, may pose unwarranted risks in administering the investigational product to the patient.
6. Uncontrolled medical condition (e.g., uncontrolled insulin-dependent diabetes mellitus).
7. Patient experiencing ongoing vomiting from any organic aetiology (including patients with history of gastric outlet obstruction or intestinal obstruction due to adhesions or volvulus), or patient with hydrocephalus.
8. Patient who experienced any vomiting, retching, or nausea within 24 h prior to the administration of the study treatment on Day 1 (Note: functional vomiting for infants, which is normally seen during the first 3 months of life, is not to be considered as vomiting).
9. Patient who received any drug with potential antiemetic effect within 24 h prior to administration of study treatment on Day 1, including but not limited to the following:

   * NK1-RAs (e.g., (fos)aprepitant or any other drug of this class)
   * 5-HT3-RAs (e.g., ondansetron, granisetron, dolasetron, tropisetron, ramosetron)
   * Benzamides (e.g., metoclopramide, alizapride)
   * Phenothiazines (e.g., prochlorperazine, promethazine, perphenazine, fluphenazine, chlorpromazine, thiethylperazine)
   * Benzodiazepines initiated 48 h prior to study treatment administration on Day 1 or expected to be administered within the efficacy assessment period, except for single doses of midazolam, temazepam, or triazolam
   * Butyrophenones (e.g., droperidol, haloperidol)
   * Anticholinergics (e.g., scopolamine, except the inhaled anticholinergics for respiratory disorders e.g., ipratropium bromide)
   * Antihistamines (e.g., diphenhydramine, cyclizine, hydroxyzine, chlorphenhyramine, dimenhydrinate, meclizine)
   * Domperidone
   * Mirtazapine
   * Olanzapine
   * Prescribed cannabinoids (e.g., tetrahydrocannabinol, nabilone)
   * Over-the-counter (OTC) antiemetics, OTC cold medications, or OTC allergy medications
   * Herbal preparations containing ephedra or ginger
10. Patient who received palonosetron within 1 week prior to administration of study treatment on Day 1.
11. Patient receiving systemic corticosteroid therapy above 0.14mg/kg or >10 mg of prednisone daily or equivalent.

    Exception:

    Dexamethasone for the prevention of CINV is permitted in association with the study treatment (Test Treatment and Reference Treatment) as per standard of care and applicable guidelines, provided its dosage is reduced by 50% in consideration of known interactions with various NK1 RAs, including fosaprepitant and fosnetupitant.
12. Patient aged <6 years who received any investigational drug (defined as a medication with no marketing authorization granted for any age or indication) within 90 days prior to Day 1, or patient aged ≥6 years who received any investigational drug within 30 days prior to Day 1, or patient any age who is expected to receive investigational drugs prior to study completion.
13. Intake of alcohol, food, or beverages (e.g., grapefruit, cranberry, pomegranate, and aloe vera juices; German chamomile) known to interfere with CYP3A4 or CYP2D6 metabolic enzymes within 1 week prior to Day 1 and during the overall study period.
14. Use of any drugs or substances known to be strong inhibitors of CYP3A4 or CYP2D6 enzymes within 1 week prior to Day 1 or planned to be used during the overall study period.
15. Use of any drugs or substances known to be CYP3A4 substrates with narrow therapeutic range within 1 week prior to Day 1 or planned to be used during the overall study period.
16. Use of any drugs or substances known to be strong inducers of CYP3A4 or CYP2D6 enzymes within 4 weeks prior to Day 1 or planned to be used during the overall study period.
17. Lactating female patient.
18. Enrolment in a previous study on netupitant (either administered alone or in combination with palonosetron).
19. Marked baseline prolongation of QTc interval (QTcF>460 millisecond [msec]). At the discretion of the investigator, criterion may be based on automatic interpretation of results.

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
COHORT 1 Neptupitant exposure parameter | From time zero ( start of IV NEPA infusion) to maximum 168 hours
  Maximum concentration (Cmax)
COHORT 1 Neptupitant exposure | From time zero ( start of IV NEPA infusion) to maximum 168 hours
  Area under the plasma concentration-time curve
COHORT 2 monitoring of AEs (safety and tolerability of IV NEPA) | Up to 31 days
  monitoring of AEs following repeated IV NEPA administration

SECONDARY OUTCOMES:
COHORT 1: To assess the PK profile of netupitant. | From Time zero ( start of IV NEPA infusion) until 168 hours
  Cmax of netupitant
COHORT 1: To assess the PK profile of fosnetupitant. | From Time zero ( start of IV NEPA infusion) until 168 hours
  Cmax of fosnetupitant
COHORT 1: To assess the PK profile palonosetron. | From Time zero ( start of IV NEPA infusion) until 168 hours
  Cmax of palonosetron
COHORT 1: To assess the PK profile of netupitant | From Time zero ( start of IV NEPA infusion) until 48 hours
  AUC0-48 of netupitant
COHORT 1: To assess the PK profile of fosnetupitant. | From Time zero ( start of IV NEPA infusion) until 48 hours
  AUC0-48 of fosnetupitant
COHORT 1: To assess the PK profile palonosetron. | From Time zero ( start of IV NEPA infusion) until 48 hours
  AUC0-48 of palonosetron
COHORT 1: To assess the PK profile of netupitant | From Time zero ( start of IV NEPA infusion) until 168 hours
  t1/2 of netupitant
COHORT 1: To assess the PK profile of palonosetron. | From Time zero ( start of IV NEPA infusion) until 168 hours
  t1/2 of palonosetron
COHORT 1 and 2: To assess the population PK profile of fosnetupitant. | From Time zero ( start of IV NEPA infusion) until 168 hours
  Clearance (CL) of fosnetupitant
COHORT 1 and 2: To assess the population PK profile of palonosetron. | From Time zero ( start of IV NEPA infusion) until 168 hours
  CL of palonosetron
COHORT 1 and 2: To assess the population PK profile of netupitant. | From Time zero ( start of IV NEPA infusion) until 168 hours
  CL/F of netupitant
COHORT 1 and 2: To assess the population PK profile of fosnetupitant | From Time zero ( start of IV NEPA infusion) until 168 hours
  Volume of compartments (V) for fosnetupitant
COHORT 1 and 2: To assess the population PK profile of palonosetron. | From Time zero ( start of IV NEPA infusion) until 168 hours
  V for palonosetron
COHORT 1 and 2: To assess the population PK profile of netupitant. | From Time zero ( start of IV NEPA infusion) until 168 hours
  V/F for netupitant

CONTACTS AND LOCATIONS:
Locations (18):
- Greece (2):
  - Aghia Sophia Children's Hospital, Pediatric Hematology/ Oncology Unit (POHemU), Athens
  - "AHEPA" University General Hospital of Thessaloniki, 2nd Department of Pediatrics, Thessaloniki
- Poland (8):
  - Department of Pediatrics, Oncology and Hematology University Children's Clinical Hospital them. Ludwik Zamenhof in Bialystok, Bialystok
  - Clinic of Pediatrics, Oncology and Hematology University Pediatric Center them M. Konopnicka SP ZOZ Central Clinical Hospital Medical University of Lodz, Lodz
  - Clinical Department of Paediatric Oncology and Haematology VOIVODSHIP SPECIALIST CHILDREN'S HOSPITAL them. prof. dr. Stanisław Popowski in Olsztyn, Olsztyn
  - Department of Pediatric Oncology, Hematology and Transplantation Clinical Hospital them. Karol Jonscher Medical University them. Karol Marcinkowski in Poznań, Poznan
  - Department of Paediatrics and Paediatric Haemato-Oncology University Clinical Hospital No. 1 them. prof. Tadeusz Sokołowski Pomeranian Medical University, Szczecin
  - Department of Paediatrics, Oncology and Paediatric Immunology, University Clinical Hospital No. 1 them. prof. Tadeusz Sokołowski Pomeranian Medical University in Szczecin, Szczecin
  - Department of Oncology and Surgical Oncology for Children and Youth Institute Mother and Child, Warsaw
  - Department of Oncology Institute "Monument - Child Health Center", Warsaw
- Romania (3):
  - Fundeni Clinical Institute, Pediatric Hematology and BMT, Bucharest
  - Oncology Institute "Prof. Dr. Al. Trestioreanu", Pediatric Oncology, Bucharest
  - Emergency Children's Hospital " Louis Turcanu, Oncology-Haematology and BMP department, Timișoara
- Turkey (Türkiye) (5):
  - Istanbul University Istanbul Faculty of Medicine Topkapı, Istanbul, Faith
  - Ankara University Faculty of Medicine Children's Hospital, Department of Children Oncology and Hematology, Ankara, Mamak
  - Erciyes University Hospitals Kanka Children's Hematology Oncology and Bone Marrow Hospital, Kayseri, Melikgazi
  - Gazi University Gazi Hospital Children Hematology and Oncology, Ankara
  - Hacettepe University Hospitals Oncology Hospital 2nd Floor Children Oncology, Ankara

IPD SHARING:
Plan to Share IPD: No
Only global trial data will be shared, not a single patient